CLINICAL TRIAL: NCT04461678
Title: Clinical Trial for Registration of HPV Nucleic Acid Genotyping Assay Kit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BDS-19CNHPV
Record Dates: First submitted 2020-06-30; First posted 2020-07-08 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening population and ASCUS referral population (Experimental): The screening population: Two cervical cytology samples will be collected from each subject. The 1st tube of SurePath liquid-based cytology sample is used for cytology test and BD Onclarity Assay HPV detection. Subjects with cytology test results ≥ ASCUS or positive HPV test results will be suggested to return for baseline colposcopy within approximately 12 weeks. In case of visible lesions under colposcopy, a biopsy of tissues at the site of the lesion will be performed; in case of no visible lesions, randombiopsy and/or ECC will be performed. Patients with histopathological results ≥ CIN2 will completed the study.
  ASCUS referral population: Female subjects with an ASCUS cytology result will be recalled undergo colposcopy, the remaining samples for cytology test collected prior to enrollment will be used for BD Onclarity Assay HPV test.
  Interventions: Diagnostic Test: HPV Genotyping Nucleic Acid Assay Kit

INTERVENTIONS:
Diagnostic Test: HPV Genotyping Nucleic Acid Assay Kit — The total sample size of screening population is approximately 12,000 cases (all females ≥ 21 years of age). Two cervical cytology samples will be collected from each subject with a tube of SurePath sample followed by a tube of PreservCyt sample. The 1st tube of SurePath liquid-based cytology sample is used for cytology test and BD Onclarity Assay HPV detection. Subjects with cytology test results ≥ ASCUS or positive HPV test results will be suggested to return for baseline colposcopy within approximately 12 weeks.

SUMMARY:
The objective of this study is to verify the clinical effectiveness of HPV Genotyping Nucleic Acid Assay Kit. This is a multi-center clinical study involving at least three study centers, each with screening sites. The protocol describes two study phases: Phase I is a baseline study of the screened population and ASCUS referral population (if necessary), the data of which will be submitted after the baseline study is completed; Phase II is a three-year follow-up study of the screened population, the data of which will be submitted again after the follow-up is completed.

DETAILED DESCRIPTION:
Baseline study of the screened population:

The total sample size of screened population is approximately 12,000 cases (all females ≥ 21 years of age). Two cervical cytology samples will be collected from each subject with a tube of SurePath sample followed by a tube of PreservCyt sample. The 1st tube of SurePath liquid-based cytology sample is used for cytology test and BD Onclarity Assay HPV detection. Subjects with cytology test results ≥ ASCUS or positive HPV test results will be suggested to return for baseline colposcopy within approximately 12 weeks. Subjects with unsatisfactory cytology results may be recalled for a second sampling 2 months after the first collection of the cervical sample. In case of visible lesions under colposcopy, a biopsy of tissues at the site of the lesion will be performed (an ECC will be performed if necessary); in case of no visible lesions, randomly biopsy and/or ECC will be performed if necessary. Patients with histopathological findings ≥ CIN2 will complete the study (see Figure 1). In the baseline colposcopy phase, if the subject is pregnant, the subject will be withdrawn from the study without colposcopy performed.

Based on the age of the subjects, different cytology results, and Surepath BD Onclarity Assay HPV results, a total of more than 500 PreservCyt samples will be selected for BD Onclarity Assay test and the HPV test for control product. For inconsistent results, a third-party sequencing method will be used to determine the final result.

SurePath sample and PreserveCyt sample collected from the same subject will be used for BD OnclarityTM Assay test to compare the consistency of test results, at least 200 samples will be enrolled only for this test. Subjects will exit the study after those HPV test without any other test.

ASCUS referral population study Female subjects with known ASCUS cytology results will be enrolled in the referral population (21-65 years old) if necessary. Female subjects with an ASCUS cytology result will be recalled to sign the informed consent to participate in the study and undergo colposcopy (within 12 weeks from the cytology sampling). For referral population, the remaining cervical samples collected prior to enrollment for cytology test will be tested with the BD Onclarity Assay HPV (see Figure 2). Such population is only used for the assessment of ASCUS triage indications and does not enter the follow-up longitudinal follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects ≥ 21 of age and < 65 of age
* Subjects who have signed the inform consent form

Exclusion Criteria:

* Pregnant subjects
* Subjects who have had cervical cytology samples taken in the last 12 months
* Subjects who have previously undergone a total hysterectomy
* Subjects who have previously undergone cone resection, LEEP, cervical laser surgery, cervical cryosurgery or uterine ablation within 3 years
* Subjects who are participating in other clinical trials of cervical disease diagnostic products

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12230 (Actual)
Dates: Start 2020-08-23 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Verification of the accuracy of nucleic acid assay | 12 weeks
  The results of HPV Assay of test product and reference product
PLR and NLR in ASCUS population | 12 weeks
  Clinical sensitivity (Sn), clinical specificity (Sp), positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio (PLR) and negative likelihood ratio (NLR) of carcinogenic HPV+ in case of ≥CIN2.
HPV risk of ≥ CIN2 in NILM 30+ population | 3 years
  1. absolute risk and 95%CI of HPV+, HPV 16 / 18/45 +, HPV31 / 33_58 / 52; HPV51 / 35_39_68 / 56_59_66 + and HPV- in case of ≥ CIN2
  2. Relative risk and 95%CI of HPV+ and HPV- in case of ≥ CIN2
  3. Relative risk and 95%CI of HPV 16 / 18/45 and HPV- in case of ≥ CIN2
  4. Relative risk and 95%CI of HPV 31 / 33_58 / 52 and HPV- in case of ≥ CIN2
  5. Relative risk and 95%CI of HPV 51, 35 / 39 / 68, 56 / 59/66 and HPV- in case of ≥ CIN2
  6. Relative risk and 95%CI of HPV 16 / 18/45 + and HPV 31 / 33_58 / 52 + in case of ≥ CIN2
  7. Relative risk and 95%CI of HPV 16 / 18/45 + and HPV 51, 35 / 39 / 68, 56 / 59/66 + in case of ≥ CIN2
  8. Relative risk and 95%CI of HPV 31 / 33_58 / 52 + and HPV 51, 35 / 39 / 68, 56 / 59/66 + in case of ≥ CIN2
HPV risk of ≥ CIN2 in Primary screening | 3 years
  1. Absolute risk and 95%CI of NILM, HPV-, HPV +, HPV16 / 18/45 +, HPV 31 / 33_58 / 52 +, HPV 51, 35 / 39 / 68, 56 / 59/66 + and HPV in case of ≥ CIN2
  2. Relative risk and 95%CI of NILM and HPV- in case of ≥ CIN2
  3. Relative risk and 95%CI of HPV+ and HPV- in case of ≥ CIN2
  4. Relative risk and 95%CI of HPV 16 / 18/45+ and HPV- in case of ≥ CIN2
  5. Relative risk and 95%CI of HPV 31 / 33_58 / 52 and HPV- in case of ≥ CIN2
  6. Relative risk and 95%CI of HPV 51, 35 / 39 / 68, 56 / 59/66 and HPV- in case of ≥ CIN2
  7. Relative risk and 95%CI of HPV 16 / 18/45 + and HPV 31 / 33_58 / 52 + in case of ≥ CIN2
  8. Relative risk and 95%CI of HPV 16 / 18/45 + and HPV 51, 35 / 39 / 68, 56 / 59/66 + in case of ≥ CIN2
  9. Relative risk and 95%CI of HPV 31 / 33_58 / 52 + and HPV 51, 35 / 39 / 68, 56 / 59/66 + in case of ≥ CIN2

CONTACTS AND LOCATIONS:
Overall Officials: Shaokai Zhang, Principal Investigator — Henan Cancer Hospital
Locations (5):
- China (5):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Obstetrics&Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Heping Hospital Affilated to Changzhi Medical College, Changzhi, Shanxi
  - Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No